CLINICAL TRIAL: NCT05883267
Title: Virtual Reality's Impact on Children With Type 1 Diabetes: a Randomized Cross-over Trial on Anxiety, Pain, Adherence, and Glycemic Control
Brief Title: Virtual Reality and Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: SHEBA-21-816421-NG-CTIL
Record Dates: First submitted 2023-04-23; First posted 2023-05-31 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2023-04

CONDITIONS: Virtual Reality

STUDY DESIGN:
Intervention Model Description: Children will be randomized to one of two interventions for diabetes management: group 1 will use VR glasses first and group 2 will listen to vocal-guided affective imagery first (audio). After 1 month, the interventions will be crossed over.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality (Experimental): The VR glasses will be PICO model neo 2. The visual and vocal data content include both calming, affective imagery and interactive gaming, supplied by "XR-Health Israel Ltd". The vocal-guided affective imagery during the procedure will be identical to the vocal guide in the VR glasses.
  Interventions: Device: Virtual reality glasses
- Audio (Active Comparator): The vocal-guided affective imagery during the procedure will be identical to the vocal guide in the VR glasses.
  Interventions: Device: Vocal-guided affective imagery

INTERVENTIONS:
Device: Virtual reality glasses — "PICO" model neo 2 VR glasses
  Arms: Virtual reality
Device: Vocal-guided affective imagery — Audio via telephone
  Arms: Audio

SUMMARY:
For children with type 1 diabetes (T1D), pain and needle phobia can cause postponing of changes in insulin pump infusion sets and continuous glucose monitors, and thus worsen glycemic control. We aim to assess the effectiveness of virtual reality (VR) technology, in reducing pain and anxiety, and improving regimen adherence and glycemic control among children with type 1 diabetes (T1D).

Children with T1D, managed with continuous glucose monitoring and insulin pumps, will be recruited for a randomized cross-over trial. Children will be randomized to one of two interventions for diabetes management: group 1 will use VR glasses first and group 2 will listen to vocal-guided affective imagery first (audio). After 1 month, the interventions will be crossed over. The outcome measures will include pain and anxiety assessment, regimen adherence, glycemic control, and patient-reported outcome measures (PROMs) of VR satisfaction and effectiveness.

DETAILED DESCRIPTION:
Children with T1D aged 8 to 15 years old, managed with CGM and insulin pumps, will be screened for participation. Key exclusion criteria include medical conditions that precluded use of the VR tool, such as epilepsy or vertigo, and diagnosed anxiety disorder.

Children will be randomly assigned (1:1 ratio) to one of the two groups. Upon every change of a CGM or pump infusion set, parents will be instructed to actively coach the child to use the designated intervention, VR glasses, or vocal-guided affective imagery, during the entire procedure. The VR glasses will be "PICO" model neo 2. The visual and vocal data content include both calming, affective imagery and interactive gaming, supplied by "XR-Health Israel Ltd". The vocal-guided affective imagery during the procedure will be identical to the vocal guide in the VR glasses. We plan 40 children in each group. The study will last for 2 months.

Questionnaires to assess anxiety and pain will be given to the children at baseline, during every CGM / pump infusion set change (every 3-14 days, depending on the device), and at one and two months after study initiation. Regimen adherence will be measured by changes in the number of insertion sites on the participants' bodies and by their willingness to change CGM / pump infusion sets themselves. Questionnaires administered at baseline, one month, and two months after the intervention will assess the use of aiding measures. Glycemic control measures that will be measured are comprised of differences between the interventions, in the percentage of time in range (TIR) 70-180 mg/dL, the percentage of time below range I (TBRI) <70 mg/dL and TBRII <54 mg/dL, the percentage of time above range I (TARI) >180 mg/dL andTARII >250 mg/dL, estimated HbA1c as measured by glucose management indicator (GMI), mean glucose, standard deviation, and the coefficient of variation (CV). A questionnaire that will assess the effectiveness and satisfaction of VR, and will evaluate the relief of diabetes distress following the intervention will be given at baseline, 1 and 2 months after the beginning.

ELIGIBILITY:
Inclusion Criteria:

• Children and young adults aged 8-15 years with type 1 diabetes with continuous glucose monitoring (CGM) and insulin pump.

Exclusion Criteria:

* Children with medical conditions not able to use virtual reality tool, such as epilepsy or vertigo.
* Children with diagnosed anxiety disorder who are treated with medications.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Pain assessment | At baseline, during every CGM/ pump infusion set change (every 3-14 days, depending on the device), and at one and two months after study initiation.
  Questionnaires to assess pain will be given to the children at baseline, during every CGM/ pump infusion set change (every 3-14 days, depending on the device), and at one and two months after study initiation. Pain scale assessment (FACES scale) will be assessed. Range of scores for the pain scale is from 0-10. A higher number meaning worse pain.
Anxiety assessment - state anxiety | At baseline, during every CGM/ pump infusion set change (every 3-14 days, depending on the device), and at one and two months after study initiation.
  Questionnaires to assess anxiety will be given to the children at baseline, during every CGM/ pump infusion set change (every 3-14 days, depending on the device), and at one and two months after study initiation. State anxiety will be assessed using the standardized Spielberger State-Trait Anxiety Inventory (STAI). State anxiety scores range from 6-24, with a higher number meaning higher anxiety.
Anxiety assessment - trait anxiety | Baseline and 2 months after the intervention
  Questionnaires to assess anxiety will be given to the children at baseline and at two months after study initiation. Trait anxiety will be assessed using the standardized Spielberger State-Trait Anxiety Inventory (STAI). Trait anxiety scores range from 20-80, a higher number meaning higher anxiety.

SECONDARY OUTCOMES:
Regimen adherence | Baseline, 1 month and 2 months after the intervention
  Regimen adherence will be measured by changes in the number of insertion sites on the participants' bodies and by their willingness to change CGM / pump infusion sets themselves. Questionnaires administered at baseline, one month, and two months after the intervention will assess the use of aiding measures.
Glycemic control measures - percentage of time in range 70-180 mg/dL | Baseline, 1 month and 2 months after the intervention
  Glycemic control measures that will be measured are comprised of differences between the interventions in the percentage of time in range 70-180 mg/dL.
Glycemic control measures - percentage of time below range <70 mg/dL | Baseline, 1 month and 2 months after the intervention
  Glycemic control measures that will be measured are comprised of differences between the interventions in the percentage of time below range <70 mg/dL.
Glycemic control measures - percentage of time below range <54 mg/dL | Baseline, 1 month and 2 months after the intervention
  Glycemic control measures that will be measured are comprised of differences between the interventions in the percentage of time below range <54 mg/dL.
Glycemic control measures - percentage of time above range I >180 mg/dL | Baseline, 1 month and 2 months after the intervention
  Glycemic control measures that will be measured are comprised of differences between the interventions in the percentage of time above range >180 mg/dL
Glycemic control measures - percentage of time above range >250 mg/dL | Baseline, 1 month and 2 months after the intervention
  Glycemic control measures that will be measured are comprised of differences between the interventions in the percentage of time above range >250 mg/dL.
Glycemic control measures - estimated HbA1c as measured by glucose management indicator (GMI) | Baseline, 1 month and 2 months after the intervention
  Glycemic control measures that will be measured are comprised of differences between the interventions in estimated HbA1c as measured by glucose management indicator (GMI).
Glycemic control measures - mean glucose | Baseline, 1 month and 2 months after the intervention
  Glycemic control measures that will be measured are comprised of differences between the interventions in mean glucose.
Glycemic control measures - standard deviation | Baseline, 1 month and 2 months after the intervention
  Glycemic control measures that will be measured are comprised of differences between the interventions in standard deviation.
Glycemic control measures - coefficient of variation (CV) | Baseline, 1 month and 2 months after the intervention
  Glycemic control measures that will be measured are comprised of differences between the interventions in coefficient of variation (CV).
VR Satisfaction and effectiveness assessment | Baseline, 1 month and 2 months after the intervention
  A questionnaire that will assess the effectiveness and satisfaction of VR, and will evaluate the relief of diabetes distress following the intervention will be given at baseline, 1 and 2 months after the beginning.

CONTACTS AND LOCATIONS:
Overall Officials: Noah Gruber, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Noah Gruber, Ramat Gan, Please Select, Israel

IPD SHARING:
Plan to Share IPD: No
Not intended

REFERENCES:
- [Derived] Gruber N, Shemesh-Iron M, Kraft E, Mitelberg K, Mauda E, Ben-Ami M, Mazor-Aronovitch K, Levy-Shraga Y, Levran N, Levek N, Zimlichman E, Pinhas-Hamiel O. Virtual reality's impact on children with type 1 diabetes: a proof-of-concept randomized cross-over trial on anxiety, pain, adherence, and glycemic control. Acta Diabetol. 2024 Feb;61(2):215-224. doi: 10.1007/s00592-023-02195-9. Epub 2023 Oct 16. PMID 37845502